CLINICAL TRIAL: NCT00152334
Title: Treatment of Idiopathic Clubfoot Utilizing Botulinum Toxin A: A New Treatment for Correction
Brief Title: Efficacy of Botox in Patients With Idiopathic Clubfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christine Alvarez, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C01-0210; W01-0057
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2017-05

CONDITIONS: Idiopathic Clubfoot (Talipes Equinovarus)
Keywords: Efficacy study; assessment of patient outcomes following treatment
MeSH Terms: conditions — Clubfoot | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botox — All patients meeting the inclusion criteria will undergo manipulation and casting until hindfoot stall is encountered. Hindfoot stall is defined as forefoot abduction to 60 degrees but persistence of hindfoot equinus. At hindfoot stall, subjects received Botox injections at 10 IU/kg into the gastrosoleus muscle complex. Following injections, subjects were recasted.

SUMMARY:
The purpose of this study was to determine the efficacy of adding Botox injection to serial manipulations and castings in patients with clubfoot. The study hypothesis was that the use of Botox in the setting of serial manipulations and castings is an effective treatment for clubfoot.

DETAILED DESCRIPTION:
All patients meeting the inclusion criteria will undergo manipulation and casting until hindfoot stall is encountered. Hindfoot stall is defined as forefoot abduction to 60 degrees but persistence of hindfoot equinus. At hindfoot stall, subjects received Botox injections at 10 IU/kg into the gastrosoleus muscle complex. Following injections, subjects were recasted.

ELIGIBILITY:
Inclusion Criteria:

1. Children presenting with idiopathic clubfoot/feet at BC Children's Hospital
2. Children ranging in age from 1 day to 2 years old at initial treatment Children who have had previous intervention for their clubfoot (methods including surgery, Ponseti method, Kite method, physical therapy method) and had a clubfoot recurrence requiring re-intervention

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2005-09; Primary Completion 2016-03 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The rate of successful clubfoot correction from a single Botox injection. This coincides with entrance into Boots and Bars. This was measured 8 weeks following injection. | 8 weeks

SECONDARY OUTCOMES:
Secondary outcomes of the study as outlined in protocol (include time of measurement) | See protocol
Secondary Outcomes: Patient outcomes collected at every patient visit including: | See protocol
1. Ankle range of motion (dorsiflexion and plantarflexion) (collected at every visit) | See protocol
2. Heel Bisector Scores (collected at every visit) | See protocol
3. Pedobarographs (every 6 months from 18 months to 5 years) | See protocol
Gait Analysis (every 2 years from 5 years of age until skeletal maturity) | See protocol

CONTACTS AND LOCATIONS:
Overall Officials: Christine Alvarez, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Department of Orthopaedics, Vancouver, British Columbia, Canada